CLINICAL TRIAL: NCT07388407
Title: Pharmacogenetics of Leflunomide in the RA Management
Brief Title: Pharmacogenetics of Leflunomide in the Management of Rheumatoid Arthritis
Status: Recruiting | Type: Observational
Sponsor: Foundation University Islamabad (Other)
Collaborators: Shifa Tameer-e-Millat University (Other)
Responsible Party: Sponsor
Other Study IDs: FUMCRCT3
Record Dates: First submitted 2026-01-02; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Rhematoid Arthritis
Keywords: RA; SNP; Leflunomide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — 5ml blood after recruitment of subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RA patients taking Leflunomide: RA patients in Pakistani population taking Leflunomide as a single DMARD
  Interventions: Drug: Study for the correlation of SNPs with efficacy and toxicity of Leflunomide in RA patients

INTERVENTIONS:
Drug: Study for the correlation of SNPs with efficacy and toxicity of Leflunomide in RA patients — Study for the correlation of SNPs with efficacy and toxicity of Leflunomide in RA patients

SUMMARY:
1. Patients taking leflunomide as the only disease-modifying anti-rheumatic drug (DMARD) will be recruited after consent.
2. Blood sample for DNA extraction will be taken The patient will be followed up till two visits 3 months apart, and efficacy and toxicity will be checked using DAS28, ultrasonography, and blood tests for ESR, CRP, anti-CCP, liver function tests, etc. The data form for toxicity will be filled.
3. DNA will be extracted in the laboratory, and SNP will be identified.
4. The efficacy and toxicity data will be studied against the SNPs found
5. An algorithm will be constructed for Pakistani RA patients taking leflunomide.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is an inflammatory autoimmune disease. Its prevalence in Pakistan is approximately 0.5% of the general population. Early introduction of disease-modifying anti-rheumatic drugs (DMARDs) along with appropriate intensification of DMARDs (the treat-to-target approach) is the most effective treatment strategy. Leflunomide, a prodrug, is a second-line DMARD used in the treatment of RA. The active metabolite of teriflunomide inhibits dihydroorotate dehydrogenase (DHODH) enzyme This prevents de novo synthesis of pyrimidines. Hence, T-cell proliferation that is characteristic of RA is inhibited. Pharmacogenetic studies specify the relationship of single nucleotide polymorphisms (SNPs) to the variability in LEF serum levels with potential relevance to effectiveness and tolerability in individual RA patients.

As a single agent in RA the efficacy of leflunomide is second line. Almost 30% of patients quit methotrexate in the first year of treatment, and leflunomide is less expensive than biologic DMARD & has fewer A/E. However, it has shown an efficacy rate of almost 68% in active RA. Trials show that 58.1% of patients experience one adverse effect due to leflunomide & 29% withdraw therapy due to them. Thus, the "Treat-to-target" approach can fail, and permanent joint damage occurs, leading to disability Thus, a prospective study of RA patients in Pakistani population taking Leflunomide as a single DMARD (with or without steroids) analyzing variations in the genes encoding DHODH and ABCG2 with outcomes of the treatment, studying both efficacy and toxicity.

Hypothesis: There is a significant relationship between DHODH, ABCG2 gene polymorphisms with clinical effects and the toxicity of leflunomide.

The aim of this study is to determine whether polymorphism in DHODH, ABCG2 genes is associated with responsiveness to leflunomide treatment in patients with RA.

OBJECTIVES To determine the frequency of genes polymorphism in DHODH, ABCG2 in Pakistani patients.

To find out the association of DHODH, ABCG2 gene polymorphisms with clinical effects of Leflunomide To find out the association of DHODH, ABCG2 gene polymorphisms with toxicity of Leflunomide To achieve this first we will prospectively study RA patients taking single DMARD Leflunomide reporting to FFH Rheumatology OPD. We will record the characteristics of efficacy and toxicity parameters at baseline, 3 months and 6 months. On their first visit consent to participate in the study and a 5ml blood sample will be obtained. DNA extraction followed by sager sequencing would be done. Finally, the genetic associations with the clinical parameters will be obtained using correlation and multivariate analysis on the latest version of SPSS.

Leflunomide is a conventional synthetic DMARD used in the treatment of RA when first line drugs fail; either they are ineffective or too toxic to be tolerated by the patient. Before switching on to biologics which are expensive and have a spectrum of adverse effects; a trial with an easily administered (orally given as opposed to biologics which must be given by infusion) and a cost-effective drug seems to be essential. However; the efficacy of leflunomide can generally be judged over a period of approximately 3-6 months, shortening time to disease suppression is crucial for improved outcomes in RA. It is thus desirable to avoid delays occasioned by use of leflunomide in patients in whom response is unlikely, since potentially more efficacious alternatives, such as biological DMARDs, are available. Genetic polymorphisms can influence drug responses through many pathways. The results of numerous studies confirm that genotype-based therapies are the most effective and may help to avoid the occurrence of major adverse events, as well as decrease the costs of treatment. Genetic variations influence the generation of active metabolites. The cytochrome P450 (CYP) system, particularly the enzyme encoded by CYP1A2, CYP2C19, activates leflunomide. The ABCG2 gene encodes the efflux pump and is studied for efficacy. The DHODH 19A>C (rs 3213422) polymorphism has been studied as a predictor of both efficacy and toxicity of leflunomide.

To date, LEF pharmacogenetics have not been studied in the Pakistani population. There is no insight into leflunomide genetics in Southeast Asia.

Based on genotyping, earlier identification of patients who are either resistant to LEF therapy or presumed at high risk of AEs can be done This would allow us to switch the therapy to another DMARD in a timely manner. This is also valuable because we can establish before even initiating the therapy A prospective study of RA patients in Pakistani population taking Leflunomide as a single DMARD (with or without steroids), analysing variations in the genes encoding DHODH, ABCG2 with outcomes of the treatment, and studying both efficacy and toxicity.

Is there any association between DHODH, ABCG2 gene polymorphisms with clinical effects and toxicity of leflunomide?

Methodology:

Study Design: Prospective, Observational, Cohort longitudinal study Setting: Fauji Foundation Hospital, Rawalpindi, laboratory settings of Shifa College of Medicine & Shifa College of Pharmaceutical Science, Islamabad.

Duration of Study: 24 months after the approval of the synopsis. Sample Size: N=120 using online sample size calculator for genetic studies; power of study is 80%, significance level of 0.05%, CI 95% Sampling Technique: Purposive Convenient sampling Inclusion criteria

1. At baseline, all patients should fulfill the revised ACR/EULAR criteria for RA10
2. Pakistani individuals
3. between ages of 20-75 years
4. New cases started on leflunomide/those already taking for less than a month and their biochemical and clinical data is available

Exclusion Criteria:

1. Patients not willing to participate/consent not given
2. Patients below the age of 20
3. Non- Pakistani origin
4. Taking another DMARD simultaneously
5. Compromised renal and hepatic functions
6. Cognitive impairment, neurological disease
7. Pregnant/ lactating patients
8. Patients having inflammatory bowel disease/ Irritable bowel syndrome
9. Patients with active infective diseases
10. Patients who fail to complete 3 months of leflunomide therapy Measurement of Efficacy DAS28-ESR (Disease activity score) Patients' global assessment of general health expressed on the visual analogue scale (VAS 0-100 mm).

Anticyclic citrullinated peptide antibody (anti-CCP), Monitoring of erosive changes of hands and feet observed on radiographs Monitoring of synovitis on Ultra sonography Measurement of Toxicity

* LFTs - hepatotoxicity
* Data collection for toxicity i. Nausea, Vomiting ii. Diarrhea iii. Stomach ache iv. Hair loss v. Weight gain vi. Rashes / eczema vii. Mucosal lesions, furunculosis, nail changes viii. BP ix. Number of infections during the treatment (UTIs, RTIs) x. Headache, Vertigo, Paraesthesia xi. Menstrual irregularities xii. Skin Infections

Data form is designed for that, which is attached. Patient Selection: Sample will be collected from patients receiving leflunomide treatment for RA The purpose & procedure will be explained. Consent to participate in the study will be recorded All patients will be assessed with the DAS28 at baseline and six and twelve weeks of treatment initiation. Adverse effects frequency and intensity will also be recorded on the data collection form Sample collection: 5ml blood will be collected in EDTA-anticoagulated tubes for extraction of DNA and sequencing End point: Patients will be classified into responders and non-responders (EULAR 2022 guidelines and DAS 28) All the biochemical markers and adverse effects will be studied Statistical Analysis: will be done on SPSS v27 Categorical variables will be presented as values and compared by using Chi-square test. A P-value of <0.05 will be statistically significant Quantitative variables will be expressed as the mean ± standard deviation (SD) and genotype-wise difference among groups will be assessed using one-way analysis of variance (ANOVA) with the post hoc Tukey multiple comparison test.

All SNPs will be studied, new SNPs will be reported DHODH haplotype, SNP s will be identified by in silico analysis Algorithm construction according to results for Pakistani population

ELIGIBILITY:
Inclusion Criteria:

* At baseline, all patients should fulfill the revised ACR/EULAR criteria for RA10
* Pakistani individuals
* between ages of 20-75 years
* New cases started on Leflunomide/ those already taking for less than a month and their biochemical and clinical data is available

Exclusion Criteria:

* Patients not willing to participate/ consent not given
* Patients below the age of 20
* Non- Pakistani origin
* Taking another DMARD simultaneously
* Compromised renal and hepatic functions
* Cognitive impairment, neurological disease
* Pregnant/ lactating patients
* Patients having inflammatory bowel disease/ Irritable bowel syndrome
* Patients with active infective diseases -Patients who fail to complete 3 months of leflunomide therapy-

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient of RA taking Leflunomide
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
DAS Score Measurement | 2 years
  The Disease Activity Score (DAS28) is calculated by assessing 28 tender/swollen joints, blood inflammatory markers (ESR or CRP), and patient global health (VAS), with scores <2.6 indicating remission and >5.1 indicating high disease activity. It is primarily computed using specialised calculators for Rheumatoid Arthritis.
  We will take this score at the start of leflunomide therapy, at three-month intervals and at 6 months. The significant outcome will be a 10% decrease from the baseline and will be correlated with the SNP identified.

SECONDARY OUTCOMES:
SNP identification in DHOD gene | 2 years
  SNPs detected from the Sanger sequencing will be tabulated against the efficacy, which is the DAS score and visual pain analogue.
  A 10% decrease in the baseline score will be considered significant improvement.
  An increase in the adverse effects like deranged LFTs, an increase in vomiting, and alopecia will be measured using ANOVA.
Measurement of Hepatotoxicity of Leflunomide | 2 years
  Baseline liver function tests will be recorded and then repeated at 3- and 6-month intervals to correlate with the genetic basis.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Muzammil Hassan Najmi, Study Director — Foundation University Islamabad
Locations (2):
- Pakistan (2):
  - Shifa International Hospital, Islamabad, Punjab Province
  - Fauji Foundation Hospital, Rawalpindi, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] The association of DHODH, CYP1A2, and ABCG2 gene polymorphism on efficacy and toxicity of leflunomide in the management of rheumatoid arthritis concentrations is associated with leflunomide cessation in rheumatoid arthritis. British Journal of Clinical Pharmacology, 81, 113-123.
- [Background] HOPKINS, A. M., WIESE, M. D., PROUDMAN, S. M., O'DOHERTY, C. E., UPTON, R. N. & FOSTER, D. J. R. 2016. Genetic polymorphism of CYP1A2 but not total or free teriflunomide 17
- [Background] HOCK, E. S., MARTYN-ST JAMES, M., WAILOO, A., SCOTT, D. L., STEVENSON, M., RAWDIN, A., SIMPSON, E. L., DRACUP, N. & YOUNG, A. 2021. Treat-to-Target Strategies in Rheumatoid Arthritis: a Systematic Review and Cost-Effectiveness Analysis. SN Comprehensive Clinical Medicine, 3, 838-854.
- [Background] GRABAR, P. B., ROZMAN, B., LOGAR, D., PRAPROTNIK, S. & DOLŽAN, V. 2009. Dihydroorotate dehydrogenase polymorphism influences the toxicity of leflunomide treatment in patients with rheumatoid arthritis. Annals of the Rheumatic Diseases, 68, 1367-1368.
- [Background] FLEISS, J. L., LEVIN, B. & PAIK, M. C. 2013. Statistical Methods for Rates and Proportions, Wiley. GAUTHIER, M. 2007. Simulation of polymer translocation through small channels: A molecular dynamics study and a new Monte Carlo approach.
- [Background] DEVARBHAVI, H., GHABRIL, M., BARNHART, H., PATIL, M., RAJ, S., GU, J., CHALASANI, N. & BONKOVSKY, H. L. 2022. Leflunomide-induced liver injury: Differences in characteristics and outcomes in Indian and US registries. Liver Int, 42, 1323-1329.
- [Background] DAVILA, L. & RANGANATHAN, P. 2011. Pharmacogenetics: implications for therapy in rheumatic diseases. Nature Reviews Rheumatology, 7, 537-550.
- [Background] BOHANEC GRABAR, P., ROZMAN, B., TOMŠIČ, M., ŠUPUT, D., LOGAR, D. & DOLŽAN, V. 2008. Genetic polymorphism of CYP1A2 and the toxicity of leflunomide treatment in rheumatoid arthritis patients. European Journal of Clinical Pharmacology, 64, 871 876.
- [Background] BOHANEC GRABAR, P., GRABNAR, I., ROZMAN, B., LOGAR, D., TOMSIC, M., SUPUT, D., TRDAN, T., PETERLIN MASIC, L., MRHAR, A. & DOLZAN, V. 2009. Investigation of the influence of CYP1A2 and CYP2C19 genetic polymorphism on 2-Cyano-3-hydroxy-N-[4 (trifluoromethyl)phenyl]-2-butenamide (A77 1726) pharmacokinetics in leflunomide treated patients with rheumatoid arthritis. Drug Metab Dispos, 37, 2061-8.
- [Background] ASLAM MM, J. F., JOHN P, FAN K-H, BHATTI A, FEINGOLD E, ET AL. 2020. A sequencing study of CTLA4 in Pakistani rheumatoid arthritis cases. PLoS ONE, 15, e 0239426. BABIKER-MOHAMED, M. H., BHANDARI, S. & RANGANATHAN, P. 2024. Pharmacogenetics of therapies in rheumatoid arthritis: An update. Best Practice & Research Clinical Rheumatology, 101974.
- [Background] ALMUTAIRI, K., NOSSENT, J., PREEN, D., KEEN, H. & INDERJEETH, C. 2021. The global prevalence of rheumatoid arthritis: a meta-analysis based on a systematic review. Rheumatology International, 41, 863-877.
- [Background] ALETAHA, D., NEOGI, T., SILMAN, A. J., FUNOVITS, J., FELSON, D. T., BINGHAM, C. O., 3RD, BIRNBAUM, N. S., BURMESTER, G. R., BYKERK, V. P., COHEN, M. D., COMBE, B., COSTENBADER, K. H., DOUGADOS, M., EMERY, P., FERRACCIOLI, G., HAZES, J. M., HOBBS, K., HUIZINGA, T. W., KAVANAUGH, A., KAY, J., KVIEN, T. K., LAING, T., MEASE, P., MÉNARD, H. A., MORELAND, L. W., NADEN, R. L., PINCUS, T., SMOLEN, J. S., STANISLAWSKA-BIERNAT, E., SYMMONS, D., TAK, P. P., UPCHURCH, K. S., VENCOVSKÝ, J., WOLFE, F. & HAWKER, G. 2010. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum, 62, 2569-81.